CLINICAL TRIAL: NCT02679209
Title: Clinical and Radiographic Evaluation of Amnion Chorion Membrane and Demineralized Bone Matrix Putty Allograft for Management of Periodontal Intrabony Defects: a Randomized Clinical Trial.
Brief Title: Evaluation of Amnion Chorion Membrane and Demineralized Bone Matrix Putty Allograft in Periodontal Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Professor of Oral Medicine and Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aminonchorion_DBM
Record Dates: First submitted 2016-02-07; First posted 2016-02-10 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone allograft (Experimental): commercially available demineralized bone matrix putty allograft will be used to fill in the defect after opening a periodontal flap
  Interventions: Biological: Demineralized bone matrix in putty form
- Amnion chorion membrane (Experimental): Amnion chorion commercially available allograft bioresorbable membrane as a guided tissue regeneration technique will be used to in the defect after opening a periodontal flap
  Interventions: Biological: Amnion chorion membrane

INTERVENTIONS:
Biological: Demineralized bone matrix in putty form — it is a type of bone graft from human cadavers.
  Other Names: DBM
  Arms: Bone allograft
Biological: Amnion chorion membrane — A bioresorbable allograft membrane for guided tissue regeneration from amnion and chorion parts of the placenta from pregnant females for guided tissue regeneration.
  Other Names: bioresorbable membrane
  Arms: Amnion chorion membrane

SUMMARY:
A clinical and radiographic evaluation of 2 regenerative techniques, bioresorbable membrane and bone allograft for management of periodontal intrabony defects.

DETAILED DESCRIPTION:
Twenty-two patients suffering from advanced chronic periodontitis were included in this randomized controlled clinical trial. Each subject contributed had two- or three-walled intrabony defects. Patients were randomly assigned into two groups; bioresorbable membrane or bone allograft. Clinical parameters were recorded at baseline and at 3 and 6 months postoperatively. Radiographic parameters were recorded at baseline and at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Severe chronic periodontitis patients.
* having at least one site with pocket depth ≥ 6 mm and clinical attachment level ≥ 5 mm, with radiographic evidence of bone loss as detected in periapical radiographs.

Exclusion Criteria:

* Pregnant women
* Having any given systemic disease
* Taking any type of medication and/or antibiotic therapy during the 3 months before the study
* Received periodontal treatment within the past 12 months Current or former smokers

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | change from Baseline at 6 months
  Change from baseline in clinical attachment level in mm in chronic periodontitis patients

SECONDARY OUTCOMES:
pocket depth | Baseline and 6 months
  Estimation of pocket depth in mm in chronic periodontitis patients at baseline and 6 months
bone defect area | Baseline and 6 months
  Estimation of bone fill defect area in mm square in chronic periodontitis patients at baseline and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Riham Hamdy, pHD, Study Chair — Associate Professor of Oral and Maxillofacial Radiology; Amr Temraz, BDs, Principal Investigator — Master student at Oral medicine and Periodontology department; Omnia Abouldahab, phD, Study Director — Professor of Oral Medicine & Periodontology, Cairo Unv.
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kothiwale SV, Anuroopa P, Gajiwala AL. A clinical and radiological evaluation of DFDBA with amniotic membrane versus bovine derived xenograft with amniotic membrane in human periodontal grade II furcation defects. Cell Tissue Bank. 2009 Nov;10(4):317-26. doi: 10.1007/s10561-009-9126-3. Epub 2009 Mar 10. PMID 19277899